CLINICAL TRIAL: NCT03929731
Title: To Determine Long-term Outcomes, Recurrence Rates, and Treatment Needs in Polypoidal Choroidal Vasculopathy(PCV)
Brief Title: Long-term Outcomes, Recurrence Rates, and Treatment Needs in Polypoidal Choroidal Vasculopathy (PCV)
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Gemmy Cheung Chui Ming, Professor, Singapore National Eye Centre
Other Study IDs: R1597/96/2018
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-04

CONDITIONS: Polypoidal Choroidal Vasculopathy
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — Fluorescein Angiography; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Polypoidal Choroidal Vasculopathy RCT: Participants will have completed the previous PCV RCTs: EVEREST II, PLANET and PCV T&E studies
  Interventions: Diagnostic Test: Indocyanine Green Angiography

INTERVENTIONS:
Diagnostic Test: Indocyanine Green Angiography — Intravenous injection of dye-indocyanine green
  Other Names: Optical Coherence Tomography-Angiography; Fundus photography; Fundus fluorescein; Optical Coherence Tomography

SUMMARY:
To determine long-term outcomes, recurrence rates, and treatment needs in Polypoidal Choroidal Vasculopathy (PCV). Specifically, to describe the long-term outcomes, recurrence rates and treatment patterns PCV patients 5 years after first presentation. This study will also evaluate whether polyp closure within the first 12 months of therapy is associated with better long-term visual outcome and will also determine the risk of disease development in the fellow eye

DETAILED DESCRIPTION:
The investigators will conduct a non-interventional, observational cohort study to assess the visual outcome of patients who have completed one of three recent randomized controlled trials in Polypoidal Choroidal Vasculopathy (PCV) EVERESTII, PLANET, PCV Treat and Extend (T&E) study. After completion of the randomized controlled trails (2 years for EVEREST II and PLANET; 1 year for T&E study), patients will be released from clinical trial protocol. At approximately 6 years (2019-2024), patients will be contacted by research coordinators and invited to attend a follow-up examination.

Study Design:

Non-interventional, observational, cohort study

Clinical coordinators will contact patients of:

* EVEREST II (2013-2015)
* PLANET (2014-2015)
* PCV T&E (2018-2019) at ~72 +/- 6 months after their initial baseline visits (2019-2024) Study Visits and Procedures Participants will only be expected to attend 1 evaluation clinic which will last approximately 3 hours

Contact of prior trial participants Participants from prior randomized control trials (EVEREST II, PLANET and PCV T&E) will be contacted by phone and invited to attend 1 post-trial evaluation clinic.

Historical Information A history will be elicited from the participant and extracted from available medical records.

Data to be collected will include: age, gender, ethnicity and race, past medical history and medications being used, as well as ocular diseases, surgeries, and treatment.

An assessment of visual related quality of life will be performed using the impact of visual impairment (IVI) questionnaire.

Testing Procedures The following procedures will be performed (using the study technique and by delegated personnel) as part of usual care, it does not need to be repeated specifically for the study if it was performed within the defined time (within 14 days prior to visit).

1. Best-corrected Visual Acuity (BCVA) will be measured using the ETDRS VA protocol following manifest refraction.
2. Optical Coherence Tomography/ OCT Angiography: OCT and OCTA will be performed. Both standard and enhanced depth imaging scans will be performed.
3. Ocular examination on each eye including slit lamp, measurement of intra-ocular pressure, lens assessment, and dilated ophthalmoscopy.
4. Fundus Photography
5. Fundus fluorescein and Indocyanine Green angiography: FFA and ICGA will be performed.

Disease characteristics of the study eye assessed by the investigator including:

* Activity of PCV based on ICGA.
* Presence of activity clinically as evidence by presence of hemorrhage, edema.
* Presence of activity as evidence by intra retinal or sub retinal fluid on OCT. The clinical data from the exit of trial to this visit will be accessed from medical records both paper- based and electronic formats.

All the data collected from this visit, data from the prior trial and the clinical course and treatment from the end of the trial to this visit will be anonymized and sent to the Singapore Eye Research Institution (SERI) for analysis. Only the principal investigator and study team at site and SERI will have access to the anonymized collected information.

ELIGIBILITY:
Inclusion Criteria:

* Participants will have completed the previous PCV RCTs: EVEREST II, PLANET and PCV T&E studies
* Are able to give consent for this follow up study

Exclusion Criteria:

* No exclusion criteria unless they do not meet the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will have completed the previous PCV RCTs: EVEREST II, PLANET and PCV T&E studies
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Long term prognostication | within 72 months
  Long term recurrence rates, correlated baseline characteristics and initial treatment strategies correlated to long term outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Singapore National Eye Centre
Locations (3):
- Singapore (3):
  - Singapore National Eye Centre, Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No